CLINICAL TRIAL: NCT03748810
Title: Head-to-head Comparison of Quadruple Combination Therapy With Empagliflozin and Dapagliflozin in Patients With Poorly Controlled Type 2 Diabetes (T2D) Despite Three Existing Oral Antidiabetic Drugs (OAD)
Brief Title: Head-to-head Comparison of Empagliflozin and Dapagliflozin
Status: Completed | Type: Observational
Sponsor: Chungbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Eu Jeong Ku, Clinical assistant professor, Chungbuk National University Hospital
Other Study IDs: SGLT2 inhibitor 2018
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Type2 Diabetes
Keywords: Empagliflozin; Dapagliflozin; Sodium-glucose cotransporter 2 inhibitors; Quadruple combination antidiabetic drugs
MeSH Terms: interventions — empagliflozin; Metformin; glimepiride; Dipeptidyl-Peptidase IV Inhibitors; dapagliflozin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Triple OADs failure: Empagliflozin or dapagliflozin as an add-on drug for inadequately controlled T2D patients who are already receiving a regimen of three distinct OADs, including metformin, glimepiride and dipeptidyl peptidase 4 (DPP4) inhibitors.
  Interventions: Drug: Empagliflozin; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin 25 mg once daily add on the background OADs for 3 years
  Other Names: Metformin; Glimepiride; DPP4 inhibitor
Drug: Dapagliflozin — Dapagliflozin 25 mg once daily add on the background OADs for 3 years
  Other Names: Metformin; Glimepiride; DPP4 inhibitor

SUMMARY:
This open-labeled, prospective, observational, 3-year, clinical study was conducted to compare the effectiveness and safety between empagliflozin (25 mg once daily) and dapagliflozin (10 mg once daily) in patients with inadequately controlled type 2 diabetes despite preexisting triple OAD combination.

DETAILED DESCRIPTION:
All participants included in this study were initially requested to initiate therapy with insulin, but they insisted on another form of OAD. When participants declined insulin injection and requested another OAD, they were not randomly assigned to each groups. It is fairly common among participants with T2D to decline insulin therapy, despite being aware of its importance and the benefits in controlling blood glucose. Their lack of willingness to use insulin is explained by their avoidance of painful injections, the potential for body weight gain and their fear of hypoglycemia. The investigators conducted a regimen consisting of four OADs, including empagliflozin or dapagliflozin, to confirm which regimen would be effective and safe.

ELIGIBILITY:
Inclusion Criteria:

* Inadequately controlled under triple OADs (metformin, glimepiride, dipeptidyl peptidase inhibitor) as evidenced by HbA1c 7.5-12%

Exclusion Criteria:

* Type 1 diabetes
* Gestational diabetes
* Diabetes due to secondary causes
* Receiving anticancer treatment
* Receiving glucocorticoids or immune-suppressants
* have been treated with sodium-glucose co-transporter 2 inhibitors for more than 7 consecutive days within 3 months before entering this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The targeted population consists of adult patients with type 2 diabetes mellitus treated in outpatient setting by specialists
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c from baseline to week 156 (3-year) | Baseline, week 156 (3-year)
  Changes in HbA1c from baseline to week 156 (3-year)
Changes in fasting plasma glucose from baseline to week 156 (3-year) | Baseline, week 156 (3-year)
  Changes in fasting plasma glucose from baseline to week 156 (3-year)

SECONDARY OUTCOMES:
Changes in HbA1c from baseline to week 104 (2-year) | Baseline, week 104 (2-year)
  Changes in HbA1c from baseline to week 104 (2-year)
Changes in HbA1c from baseline to week 52 (1-year) | Baseline, week 52 (1-year)
  Changes in HbA1c from baseline to week 52 (1-year)
Changes in HbA1c from baseline to week 24 | Baseline, Week 24
  Changes in HbA1c from baseline to week 24
Changes in fasting plasma glucose from baseline to week 12 | Baseline, Week 12
  Changes in fasting plasma glucose from baseline to week 12
Changes in fasting plasma glucose from baseline to week 24 | Baseline, Week 24
  Changes in fasting plasma glucose from baseline to week 24
Changes in fasting plasma glucose from baseline to week 56 (1-year) | Baseline, Week 56 (1-year)
  Changes in fasting plasma glucose from baseline to week 56 (1-year)
Changes in weight between baseline and week 156 (3-year) | Baseline, Week 156 (3-year)
  Changes in weight between baseline and week 156 (3-year)
Changes in weight between baseline and week 104 (2-year) | Baseline, Week 104 (2-year)
  Changes in weight between baseline and week 104 (2-year)
Changes in weight between baseline and week 52 | Baseline, Week 52
  Changes in weight between baseline and week 52
Changes in weight between baseline and week 24 | Baseline, Week 24
  Changes in weight between baseline and week 24
Changes in weight between baseline and week 12 | Baseline, Week 12
  Changes in weight between baseline and week 12
Changes in systolic blood pressure between baseline and week 156 (3-year) | Baseline, Week 156 (3-year)
  Changes in systolic blood pressure between baseline and week 156 (3-year)
Changes in systolic blood pressure between baseline and week 104 (2-year) | Baseline, Week 104 (2-year)
  Changes in systolic blood pressure between baseline and week 104 (2-year)
Changes in systolic blood pressure between baseline and week 52 | Baseline, Week 52
  Changes in systolic blood pressure between baseline and week 52
Changes in systolic blood pressure between baseline and week 24 | Baseline, Week 24
  Changes in systolic blood pressure between baseline and week 24
Changes in systolic blood pressure between baseline and week 12 | Baseline, Week 12
  Changes in systolic blood pressure between baseline and week 12
Changes in diastolic blood pressure between baseline and week 156 (3-year) | Baseline, Week 156 (3-year)
  Changes in diastolic blood pressure between baseline and week 156 (3-year)
Changes in diastolic blood pressure between baseline and week 104 (2-year) | Baseline, Week 104 (2-year)
  Changes in diastolic blood pressure between baseline and week 104 (2-year)
Changes in diastolic blood pressure between baseline and week 52 | Baseline, Week 52
  Changes in diastolic blood pressure between baseline and week 52
Changes in diastolic blood pressure between baseline and week 24 | Baseline, Week 24
  Changes in diastolic blood pressure between baseline and week 24
Changes in diastolic blood pressure between baseline and week 12 | Baseline, Week 12
  Changes in diastolic blood pressure between baseline and week 12
Changes in total cholesterol between baseline and week 156 (3-year) | Baseline, Week 156 (3-year)
  Changes in total cholesterol between baseline and week 156 (3-year)
Changes in triglyceride between baseline and week 156 (3-year) | Baseline, Week 156 (3-year)
  Changes in triglyceride between baseline and week 156 (3-year)
Changes in LDL-cholesterol between baseline and week 156 (3-year) | Baseline, Week 156 (3-year)
  Changes in LDL-cholesterol between baseline and week 156 (3-year)
Changes in HDL-cholesterol between baseline and week 156 (3-year) | Baseline, Week 156 (3-year)
  Changes in HDL-cholesterol between baseline and week 156 (3-year)
Percentage of patients with hypoglycemic episodes between baseline and week 156 (3-year) | Baseline, Week 156 (3-year)
  All episodes consistent with hypoglycemic episodes with or without a confirmatory blood glucose reading were collected
Percentage of patients with at least 1 episode of genitourinary tract infections between baseline and week 156 (3-year) | Baseline, Week 156 (3-year)
  Percentage of patients with at least 1 episode of genitourinary tract infections

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hyun Ahn, Study Chair — Chungbuk National University Hospital
Locations (1):
- Chungbuk National University Hospital, Cheonju, North Chungcheong, South Korea

REFERENCES:
- [Derived] Ku EJ, Lee DH, Jeon HJ, Oh TK. Long-term effectiveness and safety of quadruple combination therapy with empagliflozin versus dapagliflozin in patients with type 2 diabetes: 3-year prospective observational study. Diabetes Res Clin Pract. 2021 Dec;182:109123. doi: 10.1016/j.diabres.2021.109123. Epub 2021 Nov 3. PMID 34740742
- [Derived] Ku EJ, Lee DH, Jeon HJ, Oh TK. Empagliflozin versus dapagliflozin in patients with type 2 diabetes inadequately controlled with metformin, glimepiride and dipeptidyl peptide 4 inhibitors: A 52-week prospective observational study. Diabetes Res Clin Pract. 2019 May;151:65-73. doi: 10.1016/j.diabres.2019.04.008. Epub 2019 Apr 4. PMID 30954510